CLINICAL TRIAL: NCT01198977
Title: Telehealth-Based Exercise Program to Treat Fatigue in MS
Acronym: MS-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B4972-W
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; Fatigue; exercise; telemedicine; motivational interviewing; counseling; depression; physical activity
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief telephone-based counseling (Active Comparator): Telephone based counseling and instructional video
  Interventions: Behavioral: Brief telephone-based counseling
- Education Counseling (Placebo Comparator): Mailed Physical Activity information and instructional video only
  Interventions: Other: Education counseling

INTERVENTIONS:
Behavioral: Brief telephone-based counseling — Brief telephone-based counseling using Motivational Interviewing and physical activity goal setting and problem solving
  Arms: Brief telephone-based counseling
Other: Education counseling — Mailed informational video of exercise programs
  Arms: Education Counseling

SUMMARY:
This is a clinical trial examining a brief motivational intervention to improve adherence to exercise among individuals with MS to improve fatigue.

DETAILED DESCRIPTION:
This is a 2-arm single blind parallel group RCT comparing a brief telephone based motivational intervention to an informational control to improve adherence to exercise among individuals with MS. The primary outcome is improvement in fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis
* Veteran receiving services in VA VISN 20
* Fatigue
* Ability to ambulate
* cell phone or Household phone line
* Individual with multiple sclerosis verified by MS provider
* ambulatory

Exclusion Criteria:

* Current alcohol dependence or other substance dependence
* No working phone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-10; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron P Turner, PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Turner AP, Hartoonian N, Sloan AP, Benich M, Kivlahan DR, Hughes C, Hughes AJ, Haselkorn JK. Improving fatigue and depression in individuals with multiple sclerosis using telephone-administered physical activity counseling. J Consult Clin Psychol. 2016 Apr;84(4):297-309. doi: 10.1037/ccp0000086. Epub 2016 Feb 25. PMID 26913621
- [Derived] Turner AP, Hartoonian N, Hughes AJ, Arewasikporn A, Alschuler KN, Sloan AP, Ehde DM, Haselkorn JK. Physical activity and depression in MS: The mediating role of behavioral activation. Disabil Health J. 2019 Oct;12(4):635-640. doi: 10.1016/j.dhjo.2019.04.004. Epub 2019 Apr 30. PMID 31097413
- See also: VA Multiple Sclerosis Centers of Excellence web page — http://www.va.gov/MS

RESULTS

PARTICIPANT FLOW:
Groups:
- Telephone Counseling: Telephone based counseling and instructional video
  Brief telephone-based counseling: Motivational interviewing and exercise goal setting and problem solving
- Education Counseling: Exercise information and instructional video
  Informational video: Mailed video of exercise programs
Period: Overall Study
Arm/Group | Telephone Counseling | Education Counseling
Started | 31 | 33
Completed | 30 | 33
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants were individuals with MS recruited through (a) outpatient clinics at Veterans Affairs (VA) Puget Sound Health Care System, (b) targeted mailings to veterans in the VA MS National Data Repository who lived within the state of Washington, and (c) non-VA community-based MS support groups in the greater Puget Sound area.
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Counseling | Education Counseling | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 0 | 3 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (11.6) | 53.6 (13.1) | 53.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 22 | 19 | 41
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic, White | 27 | 26 | 53
  Other | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Fatigue
Description: Modified Fatigue Inventory Scale (MFIS) at baseline, 3-month, 6-month MFIS consisted of 21 items, ranging from 0 (never) to 4 (almost always). The total score was 0 to 84.
Time Frame: baseline, 3 months, 6 months
Population: Veterans with MS from Veterans Affairs (VA) Puget Sound Health Care System and civilians with MS from the greater Puget Sound area. Note: Telephone Counseling Group: 1=lost to follow-up, so analyzed 30 participants instead of 31.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Telephone Counseling: Telephone based counseling and instructional video
  Intervention of brief telephone-based counseling: Motivational interviewing and exercise goal setting and problem solving
- Education Counseling: Self-directed physical activity information and instructional video
  Informational video: Mailed video of Physical activity programs
Arm/Group | Telephone Counseling | Education Counseling
Number analyzed (Participants) | 30 | 33
units on a scale
  Baseline | 53.78 (2.67) | 49.65 (2.54)
  Month 3 | 45.76 (3.01) | 50.53 (2.86)
  Month 6 | 44.73 (2.78) | 49.70 (2.65)
Statistical Analysis 1: Comparison: Telephone Counseling vs Education Counseling; Test type: Non-Inferiority or Equivalence — Power analyses were conducted with GPower 3 evaluating the a priori sample size required to detect a medium-sized effect (f= .25, Cohen, 1988) for Group XTime interaction on primary DV. Assuming two-tailed alpha=.05 and autocorrelations between repeated measures of r=.50, adequate power (.80) to detect medium sized. Group Time effect (f=.25) would be achieved with a total sample size of 28. Given the sample size of 64, observed power more than adequate (.99); p = .013, ANOVA — Baseline and 3-month follow-up for arm 1 and arm 2
Statistical Analysis 2: Comparison: Telephone Counseling vs Education Counseling; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.005, ANOVA — Comparing baseline to 6-month follow-up
Statistical Analysis 3: Comparison: Telephone Counseling vs Education Counseling; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.010, ANOVA — The interaction effect between the two conditions across time. Baseline, 3-month, 6-month

2. Secondary Outcome: Depression
Description: Depression Module of the Patient Health Questionnaire (PHQ-9). 9-item self-report instrument designed to identify depressive symptoms consistent with criteria for major depressive episode in the Diagnostic and Statistical Manual for Mental Disorders, 4th Edition. Each item is rated over the last 2 weeks: 0 (not at all), 1 (several days), 2 (more than half the days), or 3 (nearly every day).
  Total Score for 9 items = 27.
Time Frame: baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Telephone Counseling | Education Counseling
Number analyzed (Participants) | 30 | 33
units on a scale
  Baseline | 11.38 (0.99) | 10.54 (0.95)
  Month 3 | 9.55 (1.08) | 10.86 (1.03)
  Month 6 | 7.90 (1.02) | 10.85 (0.98)
Statistical Analysis 1: Comparison: Telephone Counseling vs Education Counseling; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.009, ANOVA — Comparing depression scores for the telephone counseling and education counseling groups at 6 months
Statistical Analysis 2: Comparison: Telephone Counseling vs Education Counseling; Test type: Non-Inferiority or Equivalence — Power analyses were conducted with GPower 3 evaluating the a priori sample size required to detect a medium-sized effect (f= .25, Cohen, 1988) for Group X Time interaction on primary DV. Assuming two-tailed alpha=.05 and autocorrelations between repeated measures of r=.50, adequate power (.80) to detect medium sized. Group Time effect (f=.25) would be achieved with a total sample size of 28. Given the sample size of 64, observed power more than adequate (.99); p = .032, ANOVA — Interaction effects between the telephone counseling and education counseling groups over time (baseline, 3 months, 6 months)

3. Other Pre Specified Outcome: Physical Activity (Behavioral Target)
Description: First item of the Godin Leisure-Time Exercise Questionnaire (GLTEQ). GLTEQ asks participants to indicated the number of days per week they engaged in strenuous (e.g., running), moderate (e.g., easy bicycling), and mild (e.g., easy walking) exercise activities for periods of 15 min or more. Total weekly frequency is then calculated using an algorithm that multiplies the frequency of activities by 9 (strenuous), 5 (moderate), or 3 (mild) metabolic equivalents and sums each to produce a total level of physical activity in MET/min per week.
Time Frame: baseline, 3 months, 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Telephone Counseling | Education Counseling
Number analyzed (Participants) | 30 | 33
units on a scale
  Baseline | 16.37 (3.54) | 14.79 (3.37)
  Month 3 | 29.68 (3.72) | 19.74 (3.54)
  Month 6 | 31.06 (3.19) | 15.43 (3.04)
Statistical Analysis 1: Comparison: Telephone Counseling vs Education Counseling; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.049, ANOVA — Physical Activity Interaction effect between the Telephone Counseling and Education Counseling Group over time (baseline, 3 months, 6 months)
Statistical Analysis 2: Comparison: Telephone Counseling vs Education Counseling; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = .014, ANOVA — Comparing physical activity scores for the telephone counseling and education counseling groups at 6 months

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Telephone Counseling: Telephone based counseling and instructional video (Intervention)
  Brief telephone-based counseling: Motivational interviewing and exercise goal setting and problem solving
- Education Counseling: Exercise information and instructional video (Control)
  Informational video: Mailed video of exercise programs
Arm/Group | Telephone Counseling | Education Counseling
Serious Adverse Events (participants affected / at risk) | 3/31 | 4/33
Other Adverse Events (participants affected / at risk) | 24/31 | 18/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telephone Counseling (N=31) | Education Counseling (N=33)
car accident not related to study (Cardiac disorders) | 1 (1) | 0 (0) — ER visit for syncopal episode after accident: hypotensive and bradycardic.
MS exacerbation (Nervous system disorders) | 1 (1) | 2 (2) — Treated with IV steroids inpatient.
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fall from ladder
Overnight hospital stay - 24 hour observation of first dose of Fingolimod (Nervous system disorders) | 0 (0) | 1 (1) — MS disease modifying therapy. Requires overnight observation to new users.
Routine Overnight Inpatient Hospital Stay for MS Evaluation (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telephone Counseling (N=31) | Education Counseling (N=33)
Suicidal ideation (Psychiatric disorders) | 4 (4) | 5 (8)
Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Cut Thumb (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cut Thumb while sawing tree
Fall (Nervous system disorders) | 6 (7) | 3 (3) — Balance problems due to multiple sclerosis injuries from fall: twisted ankle, skinned hand, sore back, strained shoulder,
Increased MS Symptoms (Nervous system disorders) | 2 (2) | 0 (0)
ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Optic neuritis (Eye disorders) | 1 (1) | 0 (0) — from MS exacerbation
MS exacerbation (Nervous system disorders) | 2 (2) | 2 (2) — outpatient
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
muscle soreness from exercise (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — from having bronchitis
Numbness (Nervous system disorders) | 2 (2) | 1 (1) — MS symptom increase
slurred speech (Nervous system disorders) | 0 (0) | 1 (1) — MS symptom
Mobility (Nervous system disorders) | 1 (1) | 1 (1)
Fatigue (Nervous system disorders) | 2 (2) | 3 (3) — due to MS

LIMITATIONS AND CAVEATS:
Only ambulatory individuals were enrolled, thus high exclusion rate due to ambulation status. Outcome and mediating variables measured by validated self-report methods. A broad range of physical activity levels were included (most were low).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2009-06-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT01198977/ICF_000.pdf